CLINICAL TRIAL: NCT00737555
Title: A Phase 1b Dose-escalation Study to Evaluate the Safety and Tolerability of the Addition of the Aminopeptidase Inhibitor CHR-2797 to Paclitaxel in Patients With Advanced or Refractory Tumours
Brief Title: A Study of the Safety and Tolerability of the Addition of CHR-2797 to Paclitaxel in Patients With Advanced or Refractory Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chroma Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHR-2797-003; EudraCT# 2006-002498-35
Record Dates: First submitted 2008-08-18; First posted 2008-08-19 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Solid Tumor
Keywords: Solid tumour; Solid tumor; Pharmacokinetic; Interaction; dose escalation; cancer; paclitaxel
MeSH Terms: conditions — Neoplasms | interventions — tosedostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Once daily oral administration of CHR-2797 ( escalating dose groups) in solid tumour patients receiving paclitaxel infusion every three weeks
  Interventions: Drug: CHR-2797

INTERVENTIONS:
Drug: CHR-2797 — Oral once daily administration of capsules of CHR-2797, to determine safety and tolerability in patients being treated with paclitaxel infusion every 3 weeks for up to 18 weeks.
  Other Names: Aminopeptidase inhibitor; Proposed INN: tosedostat

SUMMARY:
The treatment of cancer often involves the use of more than one drug at the same time. In this study, patients are treated with the already marketed drug paclitaxel (administered every 3 weeks by infusion)and with the investigational drug CHR-2797 (given orally, once daily). The purpose of this study is to evaluate if it is safe to administer these two drugs together, and how well the combination is tolerated by patients. The first patients will receive a 90mg dose of CHR-2797; doses will be increased in subsequent patients, as long as they are adequately tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Signed, informed consent.
* Age > 18 years
* Histologically or cytologically documented locally advanced or metastatic solid tumour refractory to standard therapy or for which no standard therapy exists.
* Patients should have recovered from the acute adverse effects of prior therapies (excluding alopecia).
* Adequate bone marrow, hepatic and renal function including the following:
* Hb > 9g/dl (transfusion independent) or >10g/dl (transfusion permitted), absolute neutrophil count > 1.5 x 109/L, platelets ≥ 100 x 109/L;
* Total bilirubin ≤ 1.5 x upper normal limit;
* AST (SGOT), ALT (SGPT) ≤ 2.5 x upper normal limit
* Creatinine ≤1.5 x upper normal limit.
* Performance status (PS) ≤ 2 (ECOG scale).
* Estimated life-expectancy greater than 3 months.
* Female patients with reproductive potential must have a negative serum pregnancy test within 7 days prior to start of trial. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months after discontinuation of treatment.

Exclusion Criteria:

* Anti-cancer therapy including chemotherapy, radiotherapy, endocrine therapy, immunotherapy or use of other investigational agents within the 4 weeks prior to first dose of medication in this trial or within a longer period, depending on the defined characteristics of the agent e.g. 6 weeks for nitrosurea or mitomycin. Bisphosphonates for bone disease are permitted provided the doses are stable before and during the trial.
* Co-existing active infection or serious concurrent illness.
* Significant cardiovascular disease as defined by:

  * history of congestive heart failure requiring therapy;
  * history of unstable angina pectoris or myocardial infarction up to 6 months prior to trial entry;
  * presence of severe valvular heart disease;
  * presence of a ventricular arrhythmia requiring treatment.
* Any co-existing medical condition that in the investigator's judgement will
* substantially increase the risk associated with the patient's participation in the study.
* Psychiatric disorders or altered mental status precluding understanding of the
* informed consent process and/or completion of the necessary studies.
* Gastrointestinal disorders that may interfere with absorption of the study drug.
* Persistent grade II or greater toxicity from any cause.
* Patients with known brain tumours or metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurological dysfunction that would confound the evaluation of neurologic and other adverse events.
* More than 4 prior chemotherapy regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To determine the safety, tolerability, dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of CHR-2797 when administered in combination with paclitaxel. | 18 weeks

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic profile of the combination of CHR-2797 and paclitaxel and identify any pharmacokinetic interaction between the 2 agents. | After 1st and 2nd infusion of paclitaxel
To determine response and response duration, time to progressive disease or treatment failure during combination therapy and in those patients who continued beyond 18 weeks on monotherapy with CHR-2797. | Maximum duration of patient treatment ( combination followed by monotherapy) was 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Carla van Herpen, Principal Investigator — UMC St Radboud; Ferry Eskens, Principal Investigator — Erasmus MC University Medical Center
Locations (2):
- Netherlands (2):
  - UMC St Radboud, Nijmegen
  - Erasmus MC University Medical Centre- Location Centrum, Rotterdam

REFERENCES:
- See also: British Journal of Cancer 103, 1362-1368 (26 October 2010) — http://www.nature.com/bjc/journal/v103/n9/full/6605917a.html